CLINICAL TRIAL: NCT02682602
Title: In Vivo Determination of Total Hip Arthroplasty (THA) Kinematics and Sound for Subjects for Normal, Diseased and Implanted Hips
Brief Title: THA Kinematics and Sound for Subjects for Normal, Diseased and Implanted Hips
Status: Completed | Type: Observational
Sponsor: The University of Tennessee, Knoxville (Other)
Collaborators: DePuy Synthes (Industry)
Responsible Party: Principal Investigator, Richard Komistek, Fred M. Roddy Professor of Biomedical Engineering, The University of Tennessee, Knoxville
Other Study IDs: 2631FB; IIS-14002 (Other Grant/Funding Number: DePuy Synthes)
Record Dates: First submitted 2015-11-20; First posted 2016-02-15 (Estimated); Results first posted 2019-11-08 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Hip Injuries
Keywords: total hip arthroplasty
MeSH Terms: conditions — Hip Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (3):
- Diseased Hip: Subjects will have a diseased hip which requires replacement, which will be implanted with either DePuy Synthes Summit/Pinnacle total hip arthroplasty (THA) or the Corail/Pinnacle THA.
  Interventions: Radiation: Computer tomography; Radiation: Fluoroscopy surveillance
- Normal Hip: Subjects will have a normal hip.
  Interventions: Radiation: Computer tomography; Radiation: Fluoroscopy surveillance
- Implanted Group: All subjects from the Diseased Hip group were implanted with either DePuy Synthes Summit/Pinnacle total hip arthroplasty (THA) or the Corail/Pinnacle THA
  Interventions: Device: DePuy Synthes total hip arthroplasty; Radiation: Fluoroscopy surveillance

INTERVENTIONS:
Device: DePuy Synthes total hip arthroplasty
  Other Names: DePuy Synthes Summit/Pinnacle THA; DePuy Synthes Corail/Pinnacle THA
  Groups: Implanted Group
Radiation: Computer tomography — Computer tomography (CT) scan of the hip for creation of bone models.
  Groups: Diseased Hip; Normal Hip
Radiation: Fluoroscopy surveillance — Fluoroscopy evaluation of the hip during gait (level walking), chair rise, and ramp ascent and descent activities. Sound/vibration data will be collected simultaneously via non-invasive sensors attached to the hip joint.

SUMMARY:
The objective of this study is to analyze subjects having a normal hip and compare the in vivo kinematics to subjects requiring a total hip arthroplasty (THA) due to having a diseased hip and then later post-operative to their implanted hip. Ten subjects will have a normal hip, ten hips will be diseased, requiring a THA and then those ten diseased hips will be re-analyzed at least six months post-operatively after implantation of a THA.

ELIGIBILITY:
Inclusion Criteria for diseased/implanted subjects:

* Subjects will require a THA and will be implanted with either Summit/Pinnacle THA or Corail/Pinnacle THA.
* Patients must be at least six months post-operative with no other surgical procedures conducted within the past six months that will prohibit them from performing the study activities.
* Patients must be between 40-85 years of age.
* Potential subjects will have a body weight of less than 250 lbs.
* Participants must have Body Mass Index (BMI) of less than 38.
* Potential subjects' THAs should be judged clinically successful with a HHS >90.
* Subjects must have demonstrated no evidence of post-operative hip subluxation or dislocation.
* Subjects must not walk with a detectable limp and must be able to actively abduct their operated hip against gravity without difficulty.
* Participants must be able to walk on level ground, ascend and descend a ramp and rise from a chair without assistance.
* Patients from the physician's list who do not meet the study requirements will not be considered.
* Patients must be willing to sign the Informed Consent (IC)/HIPAA form to participate in the study.

Exclusion Criteria for diseased/implanted subjects:

* Pregnant, potentially pregnant or lactating females. To satisfy radiation protocol, each female subject will be asked if she is pregnant, or possibly could be pregnant. A pregnant person will not be allowed to participate in the study.
* Subjects without one of the two types of required hip implants.
* Subjects who have had surgery within the past 6 months that would prohibit them from performing level walking, ascend and descend a ramp and rise from a chair without aid or support of any kind.
* Subjects who are unable to perform level walking, ascend and descend a ramp and rise from a chair without aid or support.
* Subjects with pain, functional deficits, or generalized inflammatory.
* Subjects who walk with a detectable limp.
* Subjects who cannot actively abduct their operated hip against gravity without difficulty.
* Subjects who are unwilling to sign IC/HIPAA document.
* Subjects who have a HHS <90.

Inclusion Criteria for normal subjects:

* Patients must not have any kind of hip implant.
* Subjects must not have had any type of hip surgery or any pathological hip conditions, including osteoarthritis, or hip pain.
* Patients must be between the ages of 18 and 65.
* Potential subjects will have a body weight of less than 250 lbs.
* Participants must have BMI of less than 38.
* Pregnant or potentially pregnant females will be excluded from the study. To satisfy radiation protocol, each female subject will be asked if she is pregnant, or possibly could be pregnant. A pregnant person will not be allowed to participate in the study.
* Participants must be able to walk on level ground, ascend and descend a ramp and rise from a chair without aid of any kind or have had any kind of surgical procedure within the past 6 months that would affect his/her ability to perform the study activities.
* Patients must be willing to sign the IC and HIPAA forms to participate in the study.
* Patients must be between 160cm (5'3) and 193cm (6'4) tall

Exclusion Criteria for normal subjects:

* Pregnant, potentially pregnant or lactating females. To satisfy radiation protocol, each female subject will be asked if she is pregnant, or possibly could be pregnant. A pregnant person will not be allowed to participate in the study
* Subjects with any kind of hip implant.
* Subjects who have had any past hip surgery, have pathological hip conditions and/or hip pain.
* Subjects who have had surgery within the past 6 months that would prohibit them from performing level walking, ascend and descend a ramp and rise from a chair without aid or support of any kind.
* Subjects who are unable to perform level walking, ascend and descend a ramp and rise from a chair without aid or support.
* Subjects who are unwilling to sign IC/HIPAA document.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with a diseased hip that requires THA. OR Subjects with a normal hip.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2016-04; Primary Completion 2018-12 (Actual); Study Completion 2019-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Komistek, Ph. D., Principal Investigator — The University of Tennessee
Locations (3):
- United States (3):
  - Northside Hospital- Forsyth , GA 30041, Cumming, Georgia
  - Abercrombie Radiology, Knoxville, Tennessee
  - The University of Tennessee, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No
Researchers would like to retain this study data in our secure database so as to continue to add relevant, current data to our digital collection to help us work with manufacturers in the future to create better implants that last longer and will not require revision surgery. Participants will be asked if their study data may remain a part of the University of Tennessee's Center for Musculoskeletal Research data collection for use in future studies in the IC. Identifiers are automatically removed from the database upon entry into the secure server. Data shared with sponsors is de-identified.

RESULTS

PARTICIPANT FLOW:
Groups:
- Diseased/Implanted Hip: Subjects with a diseased hip which requires replacement, which will be implanted with either DePuy Synthes Summit/Pinnacle total hip arthroplasty (THA) or the Corail/Pinnacle THA.
- Normal Hip: Subjects with a normal hip.
Period: Pre-operative Diseased & Normal Hips
Arm/Group | Diseased/Implanted Hip | Normal Hip
Started | 11 | 10
Completed | 10 | 10
Not Completed | 1 | 0
Not completed — Unusable images | 1 | 0
Period: Post-operative Fluoroscopy for Implanted
Arm/Group | Diseased/Implanted Hip | Normal Hip
Started | 10 | 0
Completed | 7 | 0 (Nonimplanted subjects were not analyzed again for the second period, because this would be redundant)
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diseased/Implanted Hip | Normal Hip | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Categorical [Count of Participants; unit: Participants] — Population: One diseased hip subject's pre-operative data images collected from fluoroscopy were unusable and this subject did not participate in post-operative data collection, but participation in pre-operative fluoroscopy counts toward study enrollment. An additional subject was enrolled to attempt to acquire the ten data sets in the protocol.
  Participants
    number analyzed (Participants) | 10 | 10 | 20
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 6 | 5 | 11
    >=65 years | 4 | 5 | 9
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One subject's pre-operative fluoroscopy images were unusable and this subject did not participate in post-operative data collection. Participation in pre-operative fluoroscopy counts toward total study enrollment.
  Participants
    number analyzed (Participants) | 10 | 10 | 20
    Female | 4 | 5 | 9
    Male | 6 | 5 | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Population: One subject's pre-operative fluoroscopy images were unusable and this subject did not participate in post-operative data collection. This subject's participation in pre-operative data collection counts toward study enrollment.
  participants
    United States: number analyzed (Participants) | 10 | 10 | 20
    United States | 10 | 10 | 17

OUTCOME MEASURES:

1. Primary Outcome: Magnitude of Hip Separation During Primary Heel Strike
Description: Negative values indicate hip compression, position values indicate hip separation. All "Diseased Hip" subjects were re-analyzed approximately 2 years postoperatively to yield the "Implanted Hip" group.
Time Frame: Approximately 2 years postoperatively.
Population: All "Diseased Hip" subjects were re-analyzed approximately 2 years postoperatively to yield the "Implanted Hip" group.
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Diseased Hip (Baseline): Subjects with a diseased hip which requires replacement, which will be implanted with either DePuy Synthes Summit/Pinnacle total hip arthroplasty (THA) or the Corail/Pinnacle THA.
- Implanted Hip: Subjects from diseased hip group who were implanted with DePuy Synthes Summit/Pinnacle total hip arthroplasty (THA) or the Corail/Pinnacle THA.
Arm/Group | Diseased Hip (Baseline) | Normal Hip | Implanted Hip
Number analyzed (Participants) | 10 | 10 | 7
mm | -0.591 (1.582) | 0.096 (1.369) | 0.558 (0.326)

2. Primary Outcome: Magnitude of Hip Separation During Contra-lateral Toe Off
Description: as for outcome 1
Time Frame: Approximately 2 years postoperatively.
Population: All "Diseased Hip" subjects were re-analyzed approximately 2 years postoperatively to yield the "Implanted Hip" group.
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Implanted Hip: Diseased hip subjects who were implanted with DePuy Synthes Summit/Pinnacle total hip arthroplasty (THA) or the Corail/Pinnacle THA.
Arm/Group | Diseased Hip (Baseline) | Normal Hip | Implanted Hip
Number analyzed (Participants) | 10 | 10 | 7
mm | -1.051 (1.235) | -0.065 (0.986) | 1.593 (0.307)

3. Primary Outcome: Magnitude of Hip Separation During Contra-lateral Heel Strike
Description: as for outcome 1
Time Frame: Approximately 2 years postoperatively.
Population: All "Diseased Hip" subjects were re-analyzed approximately 2 years postoperatively to yield the "Implanted Hip" group.
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Implanted Hip: Diseased subjects who were implanted with DePuy Synthes Summit/Pinnacle total hip arthroplasty (THA) or the Corail/Pinnacle THA.
Arm/Group | Diseased Hip (Baseline) | Normal Hip | Implanted Hip
Number analyzed (Participants) | 10 | 10 | 7
mm | -1.019 (1.808) | -0.344 (1.518) | 0.566 (0.188)

4. Primary Outcome: Magnitude of Hip Separation During Primary Toe Off
Description: as for outcome 1
Time Frame: Approximately 2 years postoperatively.
Population: All "Diseased Hip" subjects were re-analyzed approximately 2 years postoperatively to yield the "Implanted Hip" group.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Diseased Hip (Baseline) | Normal Hip | Implanted Hip
Number analyzed (Participants) | 10 | 10 | 7
mm | -0.936 (1.243) | -0.143 (1.305) | 0.512 (0.149)

ADVERSE EVENTS:
Time Frame: approximately 2 years, 8 months
Groups:
- Implanted Group: Diseased hip subjects who were implanted with either DePuy Synthes Summit/Pinnacle total hip arthroplasty (THA) or the Corail/Pinnacle THA
Arm/Group | Diseased Hip | Normal Hip | Implanted Group
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10 | 0/7
Other Adverse Events (participants affected / at risk) | 0/11 | 0/10 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-09): https://cdn.clinicaltrials.gov/large-docs/02/NCT02682602/Prot_SAP_000.pdf